CLINICAL TRIAL: NCT03824431
Title: High Definition Endoscopy With NBI. Contribution in Patients With Non-erosive Esophagitis-pHmetric , Esophageal Motility, Histological and Immunohistochemical Associative Findings With Endoscopic Microerosions
Brief Title: High Definition Endoscopy With NBI. Contribution in Patients With Non-erosive Esophagitis
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tomas Navarro Rodriguez, Clinical Professor, University of Sao Paulo General Hospital
Other Study IDs: 39198813.4.0000.0068
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: GERD
Keywords: Gastroesophageal reflux disease; Narrow Band Imaging; High definition endoscopy; Microerosions; Esophageal biopsy; Immunohistochemistry.
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with endoscopic microerosions: ==Patients with typical symptoms of Gastroesophageal Reflux Disease(GERD):
  1- High resolution definition with NBI endoscopic findings of mucosal microerosions in distal esophagus .
  .
  Interventions: Diagnostic Test: Endoscopic esophageal biopsies
- patients without microerosions: 2- High resolution definition with NBI endoscopic without findings of mucosal microerosions in distal esophagus .
  Interventions: Diagnostic Test: Endoscopic esophageal biopsies

INTERVENTIONS:
Diagnostic Test: Endoscopic esophageal biopsies
  Other Names: esophageal manometry; esophageal phmetry; esophageal biopsies

SUMMARY:
Most patients with symptomatic gastroesophageal reflux disease (GERD) have a normal upper gastrointestinal endoscopy. Attempts have been made to define new endoscopic techniques for identification of abnormalities non detected in standard endoscopic exam. The high definition endoscopy with NBI could achieve a more detailed mucosal evaluation, allowing distal esophageal microerosions identification.

The objective was validate the presence and the meaning of distal esophageal mucosal microerosions using high definition endoscopy and NBI through esophageal biopsy in gastroesophageal reflux disease symptomatic patients and the association with GERD physiopathology.

Seventy patients were selected from the gastroenterology outpatient clinic (University of Sao Paulo Hospital) Endoscopic evaluation was sequentially performed after the pHmetry and esophageal manometry. Esophageal mucosal biopsies were obtained following established protocol for histological and immunohistochemical study.

DETAILED DESCRIPTION:
In this study the investigators focused the attention on patients with symptomatic GERD according to inclusion criteria and used high definition endoscopy with NBI in an attempt to increase the possibility of esophageal microerosion identification. The study was complemented with examinations of esophageal phmetry. During endoscopy, esophageal biopsies were obtained in patients with microerosions and controls (without microerosion). The collected material was evaluated by histopathological and immunohistochemical methods (interleukins-IL6, IL8 and IL1β) in an attempt to identify inflammatory alterations. The results of this investigation could contribute to the evaluation of microerosions as an early and significant abnormality with possible participation in the pathophysiology of GERD.

General objectives To validate the presence and clinical significance of endoscopic microerosions in patients submitted to esophageal mucosal biopsies, with typical symptoms of gastroesophageal reflux, using high definition endoscopy with (NBI), prolonged pHmetry, histopathological and immuno- histochemistry.

Specific objectives

1. Validate the presence of microerosions in the distal esophagus, as found in high-resolution endoscopy with NBI, in patients with typical symptoms of Gastroesophageal Reflux Disease.
2. Verify the association of microerosions in the distal esophagus in high-resolution endoscopy exams with NBI, with the manometric findings of esophageal perfusion manometry.
3. To observe the changes in the prolonged pHmetry in patients with microerosions in the distal esophagus through high definition endoscopy with NBI.
4. To evaluate the significance of the histological and immunohistochemical changes of tissue specimens obtained in esophageal biopsies of patients with microerosions in the distal esophagus, in high definition endoscopy with NBI.

This is a prospective, descriptive and cross-sectional study that included 90 patients, with GERD complaints. Seventy patients were selected as the object of study according to previously established inclusion and exclusion criteria. The selected patients were informed about their participation and signed an informed consent term. The histopathology and immunohistochemistry studies were carried out in the Department of Pathology of the same institution.

The study patients were evaluated after selection according to the inclusion and exclusion criteria on two occasions. On the first day, the examinations of esophageal manometry and phmetria were performed. The next day the pHmetry probe was removed and then the high definition endoscopy with NBI and the biopsies in the distal esophagus were performed. This approach facilitated patient adherence, especially in relation to logistics in performing the tests, and could represent more accurately the association of the tests performed. It was previously established that incomplete data from the exams would lead to the exclusion of the patient from the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 to 70 years
* Patients with symptoms typical of GERD, on at least two different days over a week, for a period of at least three consecutive months, and with conventional upper gastrointestinal endoscopy (UGE) without oesophageal changes, performed in the last 12 months.

Exclusion Criteria:

* Hiatal hérnia
* Ulcers of the upper digestive tract
* Drugs that interfere with the physiology of the esophagus
* Esophago-gastric surgeries
* Achalasia of the esophagus
* Esophagitis (erosive, eosinophilic, medicinal, infectious, non-erosive to conventional endoscopy)
* Esophageal stricture
* Esophageal varices
* Clinical situations that prevent more detailed evaluation of the Escamo-colunar junction during endoscopy (psychomotor-agitation, cough)
* Barrett's Esophagus
* Esophageal diverticulum
* Atrophic gastritis
* Recent use of anti-inflammatories <30 days
* Systemic inflammatory / immune systemic diseases of the gastrointestinal tract
* Recent Infectious Diseases <30 days
* BMI (Body Mass Index) > 30 kg / m2
* Pregnant women
* Smoking
* Recent use of anticoagulants
* Comorbidities that may interfere with esophageal motility
* Recent use of PPI (Proton Pump Inhibitor) <7 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from the Gastroenterology Clinic (University of Sao Paulo)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
High definition endoscopy with digital chromoscopy | 2 days
  Presence or absence of microerosions in distal esophagus.